CLINICAL TRIAL: NCT00531765
Title: Sodium Bicarbonate in Preventing Contrast Induced Nephropathy (SIPCIN): A Randomized Controlled Study
Brief Title: Sodium Bicarbonate in Preventing Contrast Induced Nephropathy
Acronym: SIPCIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Fawaz Alturki, King Faisal Specialist Hospital & Research center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RAC 2071003
Record Dates: First submitted 2007-09-17; First posted 2007-09-19 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Contrast Induced Nephropathy
Keywords: contrast-induced-nephropathy,; cardiac cath; creatinine; contrast; nephropathy
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): hydration with normal saline
  Interventions: Other: sodium bicarbonate infusion
- 2 (Experimental): hydration with sodium bicarbonate
  Interventions: Other: sodium bicarbonate infusion

INTERVENTIONS:
Other: sodium bicarbonate infusion — short infusion of sodium bicarbonate

SUMMARY:
We plan to conduct an open-label, randomized, stratified, parallel-group study to compare normal saline infusion to sodium bicarbonate infusion.

DETAILED DESCRIPTION:
We plan to conduct an open-label, randomized, stratified, parallel-group study to compare normal saline infusion to sodium bicarbonate infusion. 220 adult patients scheduled for routine cardiac catheterization will be enrolled. They will stratified according to the presence or absence of DM, or an estimated GER of less than 60 ml/hr before being block-randomized to the two groups. The incidence of CIN will be determined based on the average of two measurements of creatinine level before and 48 hours after the procedure, and an increase of 25% or 0.5 mg/dL (44.2 umol/L) or more.

ELIGIBILITY:
Inclusion Criteria:

All adult patients (18 years and above) who are scheduled for cardiac catechization and have abnormal but stable renal function will be eligible for enrollment. Abnormal renal function is defined as a creatinine level exceeding the normal range (more than 115 or 96 um/L in males and females, respectively, in KFSH&RC laboratories) or eGFR less than 60 ml/min

Exclusion Criteria:

Patients who fall under any of the following categories will be excluded:

* Acute renal failure
* Cardiogenic shock
* Emergency cardiac catheterization
* Preexisting peritoneal or hemodialysis
* Pregnancy
* Recent exposure to contrast agent within the last 3 days
* Allergy to contrast or any of the above treatment
* Renal transplant,
* Patients who received dopamine, mannitol, theophyllin or other medications known to affect renal function within one week from cardiac cath
* Pulmonary edema / congestive heart failure
* Use of N-acetylcystein
* Patents on NSAIDS who can not stop using them for 48 hrs before and 48 hrs after procedure (except Aspirin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2007-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Contrast Induced nephropathy | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Fawaz Al Turki, MD, Principal Investigator — King Faisal Specialist Hospital & Research Center
Locations (1):
- King Faisal Specialist Hospital & Research Center, Riyadh, Saudi Arabia